CLINICAL TRIAL: NCT04255303
Title: Decreasing Antibiotic Prescribing in Acute Respiratory Infections Through Implementation of Nurse Driven Clinical Decision Support
Brief Title: Decreasing Antibiotic Prescribing in Acute Respiratory Infections Through Nurse Driven Clinical Decision Support
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 19-01222; 2R01AI108680-07A1 (NIH)
Record Dates: First submitted 2020-01-09; First posted 2020-02-05 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Infection
MeSH Terms: interventions — Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iCPR group (Experimental): Clinic personnel (Providers and Nurses) will receive online training that includes: 1) an overview of the project; 2) iCPR workflows including triage; 3) CPR component review and risk categories; 4) history and physical examination components of the CPRs. The online training will be followed by in-person training to reinforce the online training and teach additional skills. In-person training sessions led by study team will last approximately 60 minutes, and consist of four basic components: 1) a review of the iCPR ARI protocol and tools; 2) on-screen walk-throughs of common scenarios employing the new tools; 3) physical examination technique practice with simulated patients; A 60-minute in-person follow-up nurse training will take place 4-6 weeks after implementation of the intervention.
  Interventions: Other: Integrated clinical prediction rule (iCPR) system (iCPR)
- Control no intervention group (No Intervention): standard care will continue as usual.

INTERVENTIONS:
Other: Integrated clinical prediction rule (iCPR) system (iCPR) — The iCPR tool consists of an electronic calculator that can be used to determine whether the patient is at low, intermediate or high risk for having the diagnosis and a bundled order set (called a "Smartset"). The iCPR tool will be made available directly within the Electronic Health Record (EHR) for Registered Nurses (RNs) who are seeing patients fall into the study categories. The iCPR tool through the use of order sets will guide the RN in the patient's care. The order set for patients at low risk for these diseases will recommend supportive care including over the counter cold remedies and pain relievers. The order set for patients at intermediate or high risk of these disease will recommend diagnostic tests (rapid strep antigen or CXR) to help determine if they have the disease. Based on the results of the diagnostic tests new order sets will recommend antibiotics or supportive care
  Arms: iCPR group

SUMMARY:
This study evaluates the effects of a novel integrated clinical prediction tool on antibiotic prescription patterns of nurses for acute respiratory infections (ARIs). The intervention is an EHR-integrated risk calculator and order set to help guide appropriate, evidence-based antibiotic prescriptions for patients presenting with ARI symptoms.

DETAILED DESCRIPTION:
The proposed project will fill a critical gap in the evidence base and answer the important question: can pivoting ARI CDS tools towards nurses overcome established implementation barriers to reducing antibiotic use? The proposal is highly innovative in three ways: It uses CDS tools to embed evidence-based risk stratification to enable nurse-led ARI management. It creates a nurse training program to support this nurse-led ARI treatment pathway. It will be evaluated and optimized using evidence-based implementation frameworks that will guide assessment of the fidelity, acceptability, adoption, cost, and sustainability of the tool. This will provide comprehensive implementation measures, formative and summative, and enable a rigorous understanding of barriers and facilitators to implementing nurse-led CDS tools for reducing antibiotic overprescribing. This study will provide much needed guidance on how to implement CDS-enabled, nurse-led ARI assessment and treatment to reduce antibiotic overprescribing.

ELIGIBILITY:
Inclusion Criteria:

Clinics:

* must be primary care and/or urgent care clinics
* should have a minimum of one registered nurse (RN) full time equivalents (FTE)

Nurses :

* be licensed to see patients and prescribed and/or recommend prescriptions for patients
* work a minimum of 0.5 FTE to ensure that they are seeing sufficient numbers of patients to maintain competency
* have access to the clinic EHR system, and use regularly as part of patient care

Patients:

* patients must have been seen at a participating clinic with a complaint of cough or sore throat.
* Ages 3-70 will be included for sore throat and ages 18-70 for cough

Exclusion Criteria:

* are unable or unwilling to provide informed consent
* are unable to participate meaningfully in an intervention that involves self-monitoring using software available in English (e.g., due to uncorrected sight impairment, illiterate, non-English-speaking, dementia)
* clinics will be excluded if phone call triage of patients with sore throat and cough is not performed by RNs
* Nurses will be excluded if they do not work with the clinic EHR as part of their workflow
* Patients with a history of chronic lung disease or immunosuppression will be excluded since the CPRs were not validated in these groups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 347 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Perceive the iCPR Tool as Useful. | Month 6
  Participants will be interviewed to measure the usefulness of the iCPR tool in prescribing appropriate antibiotics.
Change in proportion of Acute Respiratory Infection (ARI) encounters with inappropriate antibiotic prescribing | Baseline, Month 36
  The number of Acute Respiratory Infection (ARI) encounters with inappropriate antibiotic prescription will be measured pre and post-intervention using EHR reports assessing ordering of antibiotics

SECONDARY OUTCOMES:
Change in Job Satisfaction of RNs and physicians | Baseline, Month 6
  Job satisfaction/ burnout of the RNs and physicians in enrolled clinics will be measured qualitatively with interviews at baseline, 6, and 12 months after implementation
Change in Job Satisfaction of RNs and physicians | Month 6, Month 12
  Job satisfaction/ burnout of the RNs and physicians in enrolled clinics will be measured qualitatively with interviews at baseline, 6, and 12 months after implementation
Number of nurse triage encounters completed | Week 2
  Adoption of using iCPR tool will be measured by the number of nurse triage encounters completed through extracted EHR data.
Number of patients requiring repeat healthcare visits | week 2
  Adoption of using iCPR tool will be measured by the number of patients requiring repeat healthcare visits through extracted EHR data.

CONTACTS AND LOCATIONS:
Overall Officials: Devin Mann, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - NYU Langone Health, New York, New York
  - University of Utah School of Medicine, Salt Lake City, Utah
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request. Requests should be directed to devin.mann@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. The investigator who proposed to use the data.

REFERENCES:
- [Derived] Stevens ER, Xu L, Kwon J, Tasneem S, Henning N, Feldthouse D, Kim EJ, Hess R, Dauber-Decker KL, Smith PD, Halm W, Gautam-Goyal P, Feldstein DA, Mann DM. Barriers to Implementing Registered Nurse-Driven Clinical Decision Support for Antibiotic Stewardship: Retrospective Case Study. JMIR Form Res. 2024 May 23;8:e54996. doi: 10.2196/54996. PMID 38781006
- [Derived] Stevens ER, Agbakoba R, Mann DM, Hess R, Richardson SI, McGinn T, Smith PD, Halm W, Mundt MP, Dauber-Decker KL, Jones SA, Feldthouse DM, Kim EJ, Feldstein DA. Reducing prescribing of antibiotics for acute respiratory infections using a frontline nurse-led EHR-Integrated clinical decision support tool: protocol for a stepped wedge randomized control trial. BMC Med Inform Decis Mak. 2023 Nov 14;23(1):260. doi: 10.1186/s12911-023-02368-0. PMID 37964232

DOCUMENTS (1):
  • Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/03/NCT04255303/ICF_000.pdf